CLINICAL TRIAL: NCT06927180
Title: SHR-A1811 Plus Pertuzumab in Combination With or Without Albumin-paclitaxel as Neoadjuvant Treatment for Early or Locally Advanced HER2-positive Breast Cancer：A Prospective, Randomized, Open-label, Phase II Trial.
Brief Title: SHR-A1811 Plus Pertuzumab in the Neoadjuvant Treatment of HER2 Positive BC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Zhenzhen Liu, Professor, Henan Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-543
Record Dates: First submitted 2025-03-04; First posted 2025-04-15 (Actual); Last update posted 2025-06-23 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer Early Stage Breast Cancer (Stage 1-3)
Keywords: Breast Cancer; HER2-positive Breast Cancer; pathologic complete response; SHR-A1811; Pertuzumab; Albumin-Paclitaxel
MeSH Terms: conditions — Breast Neoplasms; Pathologic Complete Response | interventions — pertuzumab; Docetaxel; Carboplatin; Trastuzumab

STUDY DESIGN:
Intervention Model Description: Patients who meet the inclusion criteria were randomly divided into SHR-A1811+pertuzumab and SHR-A1811+pertuzumab+albumin-paclitaxel and TCbHP group in a 1:1:1 ratio.
Masking Description: Non
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1：SHR-A1811+Pertuzumab (Experimental): Participants will receive SHR-A1811+Pertuzumab for 6 cycles.
  Interventions: Drug: SHR-A1811; Drug: Pertuzumab
- Cohort 2：SHR-A1811+Pertuzumab+Albumin-Paclitaxel (Experimental): Participants will receive SHR-A1811+Pertuzumab+Albumin-Paclitaxel for 6 cycles.
  Interventions: Drug: SHR-A1811; Drug: Pertuzumab; Drug: Albumin-Paclitaxel
- Cohort 3：TCbHP (Active Comparator): Participants will receive Docetaxel +Carboplatin +Trastuzumab +Pertuzumab for 6 cycles.
  Interventions: Drug: Pertuzumab; Drug: Docetaxel; Drug: Carboplatin; Drug: Trastuzumab

INTERVENTIONS:
Drug: SHR-A1811 — an anti-HER2 antibody-drug conjugate (ADC)
  Arms: Cohort 1：SHR-A1811+Pertuzumab; Cohort 2：SHR-A1811+Pertuzumab+Albumin-Paclitaxel
Drug: Pertuzumab — Pertuzumab
Drug: Albumin-Paclitaxel — Nab paclitaxel
  Arms: Cohort 2：SHR-A1811+Pertuzumab+Albumin-Paclitaxel
Drug: Docetaxel — Docetaxel
  Arms: Cohort 3：TCbHP
Drug: Carboplatin — Carboplatin
  Arms: Cohort 3：TCbHP
Drug: Trastuzumab — Trastuzumab
  Arms: Cohort 3：TCbHP

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of SHR-A1811 plus pertuzumab in combination with or without albumin-paclitaxel neoadjuvant therapy for early or locally advanced HER2-positive breast cancer. The main questions it aims to answer are:

* Does the pCR of SHR-A1811 plus pertuzumab with or without albumin-paclitaxel improve compared to the current standard of treatment?
* Is the safety of SHR-A1811 plus pertuzumab with or without albumin-paclitaxel better compared to the current standard of treatment? Researchers will compare SHR-A1811+pertuzumab or SHR-A1811+pertuzumab+albumin-paclitaxel to TCbHP to see if SHR-A1811 plus pertuzumab with or without albumin-paclitaxel works to treat early or locally advanced HER2-positive breast cancer.

Subjects will be randomly assigned 1:1:1 to：

* cohort 1：SHR-A1811 combined with pertuzumab for 6 cycles;
* cohort 2：SHR-A1811 combined with pertuzumab and albumin-paclitaxel for 6 cycles;
* cohort 3：TCbHP (docetaxel, carboplatin, trastuzumab and pertuzumab) for 6 cycles.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic and may require frequent medical assessments, blood tests, questionnaires, and scans.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-70 years old, ECOG 0-1 point.
* Clinical T2-T4, with any LN, M0.
* HER2+, invasive breast cancer confirmed by histopathology;(HER2 positive expression means that there is at least one case of tumor cell immunohistochemical staining intensity of 3+or positive confirmed by fluorescence in situ hybridization [FISH] in the pathological test/review of the primary focus conducted by the Pathology Department of the Research Center Hospital).
* Having clinically measurable lesions: measurable lesions displayed on ultrasound, mammography, or MR (optional) within the first month of randomization.
* Organ and bone marrow function tests within one month before chemotherapy indicate no contraindications to chemotherapy：Absolute value of neutrophil count ≥ 1.5 × 10^9/L; Hemoglobin ≥ 90g/L; Platelet count ≥ 100 × 10^9/L; Total bilirubin≤1.5 ULN (upper limit of normal value); Creatinine≤1.5 × ULN; AST/ALT ≤ 2.5 × ULN.
* Cardiac ultrasound: Left ventricular ejection fraction (LVEF ≥ 50%).
* Women of childbearing age tested negative for serum pregnancy test 7 days before randomization.
* Sign an informed consent form.

Exclusion Criteria:

* Stage IV (metastatic) breast cancer.
* Has received chemotherapy, endocrine therapy, targeted therapy, reflex therapy, etc. for this disease.
* The patient has a second primary malignant tumor, except for fully treated skin cancer.
* The patient had undergone major surgical procedures unrelated to breast cancer within 4 weeks before enrollment, or the patient has not fully recovered from such surgical procedures.
* The presence of uncontrolled cardiovascular and cerebrovascular disease, including (but not limited to) any of the following within the 6 months prior to the first dose: congestive heart failure (NYHA III or IV), myocardial infarction or cerebral infarction, pulmonary embolism, unstable angina, or arrhythmia requiring treatment at the time of screening; Primary cardiomyopathy (e.g., dilated cardiomyopathy, hypertrophic cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy, restricted cardiomyopathy, undefined cardiomyopathy); A clinically significant history of prolonged QTc, grade II type II atrioventricular block or grade III atrioventricular block or QTc interphase (F method) > 470 msec (female); Atrial fibrillation (EHRA grade ≥2b); Unmanageable hypertension, which the investigators judged unsuitable for study participation.
* Due to serious and uncontrollable other medical diseases, researchers believe that there are contraindications to chemotherapy.
* Individuals with a known history of allergies to the drug components of this protocol;
* Having a history of immunodeficiency, including HIV testing positive, or suffering from other acquired or congenital immunodeficiency diseases, or having a history of organ transplantation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2029-05-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate (pCR rate) | After surgery（within 1 month）
  After neoadjuvant chemotherapy and surgery, the resected specimen (breast + axilla) was free of any invasive cancer (ie, ypT0/is, ypN0)

SECONDARY OUTCOMES:
Invasive Disease Free Survival of 5 years | 5-year
  5-year Invasive Disease-Free Survival was defined as patients who did not experience regional, contralateral or distant recurrence, or dies during a follow-up period of at least 5 years from the date of surgery.
Event-Free Survival of 5 years | 5-year
  5-year Event-Free Survival was defined as patients who did not experience disease progression during neoadjuvant therapy, local or distant recurrence, second primary malignancy (breast or other cancer), or dies during a follow-up period of at least 5 years after treatment.
Objective Response Rate (ORR) | During neoadjuvant therapy before surgery（within 6 months）
  ORR is the proportion of patients whose tumors have shrunk significantly over the course of treatment. Specifically, ORR includes both partial response (PR) and complete response (CR). Partial response (PR) : The maximum diameter or volume of the tumor is reduced by at least 30%, but it does not completely disappear. Complete response (CR) : The tumor disappears completely and no visible signs of cancer are confirmed by imaging tests, such as CT scans, MRI, or ultrasound.
Adverse Events rate | 2-year
  Evaluate the nature, incidence and severity of chemotherapy adverse events according to CTCAE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Zhenzhen Liu, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No